CLINICAL TRIAL: NCT02245516
Title: An Exploratory, Multi-Center, Randomized, Single-Masked Study Evaluating the Effect of KPI-121 on Intraretinal or Subretinal Fluid Secondary to Retinal Vein Occlusion or Diabetic Macular Edema
Brief Title: Exploratory Study of KPI-121 Effect on Intra- or Subretinal Fluid Due to Retinal Vein Occlusion/Diabetic Macular Edema
Acronym: Molokini
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KPI-121-C-004
Record Dates: First submitted 2014-09-04; First posted 2014-09-19 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Retinal Vein Occlusion; Diabetic Macular Edema
Keywords: Intraretinal Fluid; Subretinal Fluid; Retinal Vein Occlusion; Diabetic Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- KPI-121 0.25% Ophthalmic Suspension (Active Comparator): KPI-121 0.25% Ophthalmic Suspension dosed QID for 4 weeks in subjects with Retinal Vein Occlusion or Diabetic Macular Edema
  Interventions: Drug: KPI-121 0.25% Ophthalmic Suspension
- KPI-121 1.0% Ophthalmic Suspension (Active Comparator): KPI-121 1.0% Ophthalmic Suspension dosed QID for 4 weeks in subjects with Retinal Vein Occlusion or Diabetic Macular Edema
  Interventions: Drug: KPI-121 1.0% Ophthalmic Suspension

INTERVENTIONS:
Drug: KPI-121 0.25% Ophthalmic Suspension — KPI-121 drug product will be supplied a 0.25% loteprednol etabonate as a suspension packaged opaque dropper bottles. KPI-121 drug product is a sterile, aqueous, submicron suspension of loteprednol etabonate.
  Other Names: Loteprednol etabonate 0.25%
  Arms: KPI-121 0.25% Ophthalmic Suspension
Drug: KPI-121 1.0% Ophthalmic Suspension — KPI-121 drug product will be supplied a 1.0% loteprednol etabonate as a suspension packaged opaque dropper bottles. KPI-121 drug product is a sterile, aqueous, submicron suspension of loteprednol etabonate.
  Other Names: Loteprednol etabonate 1.0%
  Arms: KPI-121 1.0% Ophthalmic Suspension

SUMMARY:
The primary objectives of the study are to evaluate the safety and effect of KPI-121 0.25% ophthalmic suspension and KPI-121 1.0% ophthalmic suspension on intraretinal or subretinal fluid secondary to Retinal Vein Occlusion or Diabetic Macular Edema.

DETAILED DESCRIPTION:
This is a multicenter, randomized, single-masked study evaluating the safety and effect of topical ocular administration of either KPI-121 0.25% ophthalmic suspension or KPI-121 1.0% ophthalmic suspension in subjects with intraretinal or subretinal fluid secondary to Retinal Vein Occlusion or Diabetic Macular Edema.

ELIGIBILITY:
Inclusion Criteria:

* Have documented presence of intraretinal or subretinal fluid secondary to Retinal Vein Occlusion or Diabetic Macular Edema at Screening

Exclusion Criteria:

* Treatment with topical, intravitreal injection, posterior sub-Tenon's, or periocular corticosteroids within 120 days prior to Visit 1 and for the duration of the study
* History of uncontrolled glaucoma, IOP over 21 mmHg at Visit 1, or are being treated for glaucoma in the study eye
* Any significant ocular disease that could compromise vision in the study eye (including ongoing ocular infection, wet age-related macular degeneration, myopic degeneration with active subfoveal choroidal neovascularization)
* Known hypersensitivity or contraindication to the investigational product(s) or their components
* Diagnosis of severe/serious ocular condition that in the judgment of the Investigator could confound study assessments or limit compliance; or severe/serious systemic disease or uncontrolled medical condition that in the judgment of the Investigator could confound study assessments or limit compliance
* Exposed to an investigational drug within 30 days prior to Visit 1 and for the duration of the study
* In the opinion of the Investigator or study coordinator, an unwillingness or inability to comply with the study protocol or inability to successfully instill eye drops

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KPI-121 1.0% Ophthalmic Suspension | KPI-121 0.25% Ophthalmic Suspension
Started | 9 | 7
Completed | 9 | 4
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KPI-121 1.0% Ophthalmic Suspension | KPI-121 0.25% Ophthalmic Suspension | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 63.2 (12.93) | 65.4 (10.34) | 64.2 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS)
Description: Best Corrected Visual Acuity (BCVA) was measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score starting at 4 meters. More letters read correctly results in a higher letter score, which represents better visual acuity.
Time Frame: Day 1 to Day 57
Population: Intent to treat- all subjects randomized
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | KPI-121 1.0% Ophthalmic Suspension | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 9 | 7
ETDRS letters | -0.9 (7.83) | -2.0 (2.00)

2. Primary Outcome: Macular Volume by SD-OCT
Description: Change in measurement (in microns) in macular volume as measured by Spectral Domain Optical Coherence Tomography (OCT)
Time Frame: Day 1 to Day 57
Population: Intent to Treat (all randomized subjects) minus subjects in each treatment group that discontinued the study prior to this time point or otherwise did not have this assessment completed
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | KPI-121 1.0% Ophthalmic Suspension | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 9 | 4
mm^3 | -0.237 (1.1607) | -0.377 (0.8190)

3. Primary Outcome: Center Subfield Retinal Thickness by SD-OCT
Description: Change in measurement (in microns) in the central subfield retinal thickness as measured by Spectral Domain Optical Coherence Tomography (OCT)
Time Frame: Day 1 to Day 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | KPI-121 1.0% Ophthalmic Suspension | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 9 | 4
micrometers (μm) | -8.2 (52.37) | 4.8 (13.99)

4. Primary Outcome: Investigator's Assessment of Leakage on the Fluorescein Angiogram
Description: Change in leakage by investigator's assessment of the fluorescein angiogram
Time Frame: Day 1 to Day 57
Population: Unable to analyze the FA data for efficacy. The efficacy variable defined in the protocol was the mean change from baseline in total area of fluorescein leakage and unfortunately the total area was not collected during the study.
Arm/Group | KPI-121 1.0% Ophthalmic Suspension | KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a subjects signed the informed consent until they exited the study at the end of Visit 5 (up to 57 days).
Arm/Group | KPI-121 1.0% Ophthalmic Suspension | KPI-121 0.25% Ophthalmic Suspension
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/7
Other Adverse Events (participants affected / at risk) | 3/9 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KPI-121 1.0% Ophthalmic Suspension (N=9) | KPI-121 0.25% Ophthalmic Suspension (N=7)
generalized weakness (General disorders) | 0 | 1 — 1 Subject had a non-ocular SAE hospitalization of generalized weakness starting on Day 7 resolved Day 28. It was mild in severity, was not considered by the Investigator to be related to study treatment and the subject discontinued from the trial.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 1.0% Ophthalmic Suspension (N=9) | KPI-121 0.25% Ophthalmic Suspension (N=7)
Increase in floaters (Eye disorders) | 1 (1) | 0 (0)
Pain (Eye disorders) | 1 (1) | 0 (0)
Punctate Epithelial Erosions (Eye disorders) | 1 (1) | 0 (0)
generalized weakness (General disorders) | 0 (0) | 1 (1)
Soreness (Eye disorders) | 0 (0) | 1 (1)
Worsening of Hypercholesterolemia (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No submission for publication or public disclosure will be made by the PI until after the publication of the results of the multi-center clinical trial by the Sponsor. Thereafter, PI shall provide KALA with an advance copy of any proposed publication or public disclosure at least sixty (60) days prior to the planned date of submission or disclosure and KALA shall have forty-five (45) days from the date of its receipt to recommend changes.